CLINICAL TRIAL: NCT06569355
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of VCT220 Tablets in Overweight/Obese Subjects
Brief Title: A Study to Evaluate the Efficacy and Safety of VCT220 in Obesity Chinese Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vincentage Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VCT220-II-02
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-08

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 80mg dose group (Experimental): Participants will receive VCT220 or placebo tables in 2 weeks dose titration period and take the maintanance dose 80 mg from week 3 to week 16.
  Interventions: Drug: VCT220; Drug: Placebo
- 120mg dose group (Experimental): Participants will receive VCT220 or placebo tables in 4 weeks dose titration period and take the maintanance dose 120 mg from week 5 to week 16.
  Interventions: Drug: VCT220; Drug: Placebo
- 160mg dose group fast titration (Experimental): Participants will receive VCT220 or placebo tables in 4 weeks dose titration period and take the maintanance dose 160 mg from week 5 to week 16.
  Interventions: Drug: VCT220; Drug: Placebo
- 160mg dose group slow titration (Experimental): Participants will receive VCT220 or placebo tables in 6 weeks dose titration period and take the maintanance dose 160 mg from week 7 to week 16.
  Interventions: Drug: VCT220; Drug: Placebo

INTERVENTIONS:
Drug: VCT220 — A small molecule GLP-1R agonist tablet, orally administration, once daily
Drug: Placebo — Placebo tablet

SUMMARY:
The goal of the study is to assess how VCT220 tablets affect the bodyweight when used once daily in obese or overweight adult participants

Qualified participants will be randomly assigned to one of four groups using a computerized system. Participants will get VCT220 or placebo tablets for 16 weeks and will need to take tablets each morning.

Participants will have 7 clinic visits and a final follow-up visit approximately 14 days after the last study intervention administration.

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18-75 years (inclusive) when signing the informed consent form;
2. Body mass index (BMI) ≥ 28 kg/m2 with or without concomitant diseases; or BMI ≥ 24 kg/m2 and < 28 kg/m2 combined with at least one of the following concomitant diseases: pre-diabetes (impaired fasting glucose and/or reduced glucose tolerance), hypertension, dyslipidemia, fatty liver, and obstructive sleep apnea syndrome caused by overweight (see Appendix 1 for specific definitions);
3. Subjects who have undergone diet control or exercise control alone for at least 12 weeks before screening, resulting in a stable weight within 12 weeks before screening (weight change < 5%, weight change = [maximum weight - minimum weight]/maximum weight; based on subjects' self-report);
4. Subjects who have no fertility plan and voluntarily take effective contraceptive measures without any plans to donate sperm or eggs during the study and within 90 days after the end of study;
5. Subjects who are willing and able to maintain a stable diet and exercise during the study and fill in diary cards on time; 6）Subjects who are able to understand the procedures and methods of this study, willing to complete this study in strict accordance with the clinical study protocol, and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Subjects with previously diagnosed obesity caused by endocrine diseases or single gene mutations, including but not limited to hypothalamic obesity, pituitary obesity, hypothyroid obesity, Cushing's syndrome, islet cell tumor, acromegaly, and hypogonadism;
2. Subjects who have received bariatric surgery or treatment (except for acupuncture for weight loss, liposuction, and abdominal fat removal more than 1 year from the screening period), or plan to receive bariatric surgery to treat obesity during the study, e.g., gastric bypass surgery and gastric banding;
3. Subjects who are on a weight loss program at screening and are not in the maintenance period (based on subjects' self-report);
4. Subjects who have previously been diagnosed with type 1 diabetes mellitus, type 2 diabetes mellitus, or other special types of diabetes;
5. Subjects who have used any GLP-1 receptor agonist (GLP-1RA), GLP-1 related multi-target agonist (e.g., GLP 1/glucose-dependent insulinotropic polypeptide [GIP] dual agonist and GLP 1/glucagon receptor [GCGR] dual agonist), or compound preparations containing GLP 1 agonist;
6. Subjects who have received any of the following medications or therapies within 12 weeks before screening:

   * Oral or injectable hypoglycemic medications such as dipeptidyl peptidase-4 (DPP-4) inhibitors, sodium glucose cotransporter 2 (SGLT-2) inhibitors, metformin, insulin secretagogues, thiazolidinediones (TZDs), and insulin;
   * Any approved or unapproved weight loss drugs (such as orlistat, lorcaserin, phentermine/topiramate, and naltrexone/bupropion) or Chinese herbal medicines, health care products, meal replacements, etc., affecting body weight;
   * Use of any drugs that might significantly change body weights, including systemic (i.e., intravenous, oral, or intra-articular administration) glucocorticoids for more than 1 week; tricyclic antidepressants; antipsychotic or antiepileptic drugs (e.g., imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine hydrochloride, clozapine, olanzapine, valeric acid and its derivatives, lithium preparations, and thioridazine), etc.;
7. Subjects who meet any of the following criteria related to cardiac function:

   * History of myocardial infarction, coronary angioplasty or bypass graft, heart valve disorders or cardiac valve prostheses, clinically significant unstable arrhythmia, unstable angina, transient ischemic attack, cerebrovascular accident, etc., within 6 months before screening;
   * Class III or IV congestive cardiac failure according to New York Heart Association (NYHA) classification;
   * Subjects with serious arrhythmia requiring treatment (such as long QT syndrome) and not suitable for the clinical study as assessed by the investigator;
   * Poorly controlled hypertension before screening (i.e., systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg);
   * Presence of clinical abnormalities (e.g., QTcF > 450 msec, complete left bundle branch block, signs of acute or unexplained myocardial infarction, ST-segment changes suggestive of myocardial ischemia, second or third degree atrioventricular block, or serious bradyarrhythmia or tachyarrhythmia) by electrocardiography (ECG) at screening that might affect the safety of subjects or the interpretation of study results;
   * Resting heart rate > 100 beats/min;
   * Other cardiac function abnormalities with clinical significance judged by the investigator;
8. Currently with thyroid dysfunction that is not well controlled with a stable dose of medications, or with clinically significant abnormalities noted in thyroid function test results at screening;
9. History of medullary thyroid cancer, multiple endocrine neoplasia (MEN) syndrome type 2A or 2B or relevant family history (family history is defined as diseases in a first-degree relatives);
10. Subjects diagnosed with malignancies within 5 years before screening (except for cured cutaneous basal cell carcinoma or cervical carcinoma in situ);
11. History of acute or chronic pancreatitis, symptomatic gallbladder disease (such as multiple gallstones), pancreatic injury, and other high-risk factors that may lead to pancreatitis;
12. Subjects with clinically significant abnormal gastric emptying (such as gastric outlet obstruction), severe chronic gastrointestinal diseases (active ulcer within 6 months), long-term use of drugs with direct effects on gastrointestinal motility (including but not limited to mosapride, cisapride, etc.), or gastrointestinal surgery (except for polypectomy and appendectomy) within 6 months before screening, who are not suitable for the clinical study as assessed by the investigator;
13. History of organ transplantation, or previous or current serious autoimmune diseases;
14. Subjects who have a history of major surgery within 6 months before screening, or plan to undergo surgery that might affect study completion or compliance;
15. Subjects with a history of moderate to severe depression and anxiety, or a history of serious mental illness, or a depression screening scale (PHQ-9) score ≥ 15 at screening;
16. Subjects with previous suicidal tendency or suicidal behavior;
17. Subjects with any laboratory test parameter meeting any of the following criteria at screening:

    * Glycosylated hemoglobin (HbA1c) ≥ 6.5%;
    * Fasting plasma glucose (FPG) ≥ 7.0 mmol/L;
    * Glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 as calculated using the CKD-EPI formula;
    * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥ 3.0 × upper limit of normal (ULN);
    * Total bilirubin (TBIL) > 1.5 × ULN;
    * Blood amylase or blood lipase > 1.5 × ULN;
    * Fasting triglycerides (TG) > 5.7 mmol/L;
    * Fasting C-peptide < 0.8 ng/mL (or < 0.26 nmol/L);
    * Calcitonin ≥ 1.0 × ULN;
    * Hemoglobin (Hb) < 110 g/L (males) or < 100 g/L (females);
18. Subjects who are positive for hepatitis B virus surface antigen (HBsAg) (except for those with hepatitis B virus deoxyribonucleic acid [HBV-DNA] quantitative results lower than the lower limit of reference range and not using anti-hepatitis B virus drugs at screening), receiving anti-hepatitis B virus drugs, positive for hepatitis C virus (HCV) antibody, positive for human immunodeficiency virus (HIV) antibody, or positive for treponema pallidum antibody (Tp-Ab) at screening;
19. Subjects with known allergies to GLP-1 receptor agonists or relevant excipients;
20. Subjects who have previously participated in weight loss clinical trials; those who have participated in any clinical trial for drug or medical device (except for weight loss clinical trials) as subjects within 12 weeks before screening, or subjects who have participated in any clinical trials in which the last dose is within 5 half-lives of the investigational product before screening (whichever is longer) (such restrictions are not applicable to the subjects who fail the screening);
21. Subjects who have donated or lost ≥ 400 mL of blood or have received blood transfusion within 12 weeks before screening;
22. Subjects with a known or suspected history of alcohol or tobacco addiction, or drug abuse at screening;
23. Pregnant or lactating women;
24. Subjects with positive blood pregnancy test results at screening or before randomization (for female subjects of childbearing potential only); 25）Other conditions that make the subject unsuitable for the study as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-07-13 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Percentage change in body weight | From baseline (week 1) to week 16
  percentage-point

SECONDARY OUTCOMES:
Proportion of subjects with weight decrease ≥ 5% | From baseline (week 1) to week 16
  percentage-point
Absolute change in body weight | From baseline (week 1) to week 16
  measured in kg
Absolute change in body mass index (BMI) | From baseline (week 1) to week 16
  measured in kg/m^2
Absolute change in waist circumference | From baseline (week 1) to week 16
  measured in cm
Change in blood lipid profiles (TC, TG, LDL-C, and HDL-C) | From baseline (week 1) to week 16
  measured in mmol/L
Change in fasting plasma glucose (FPG) | From baseline (week 1) to week 16
  measured in mmol/L
Change in HbA1c (glycated haemoglobin) | From baseline (week 1) to week 16
  percentage-point
Change in fasting insulin | From baseline (week 1) to week 16
  measured in μIU/mL
Change in fasting C-peptide | From baseline (week 1) to week 16
  measured in ng/ml

OTHER OUTCOMES:
Adverse events, including treatment-emergent adverse events (TEAEs), serious adverse events (SAEs) | From baseline (week 1) to week 18
  Count of events
PK analysis-Minimum concentration | From week 1 to week 12
  measured in ng/ml
PK analysis-Maximum concentration | From week 1 to week 12
  measured in ng/ml
PK analysis-Time to maximum concentration | From week 1 to week 12
  measured in hour
PK analysis-Area under the concentration-time curve | From week 1 to week 12
  measured in h∙ng/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No